CLINICAL TRIAL: NCT02723539
Title: A Phase 1b/2a Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Efficacy of Adjunctive Treatment With Topically Applied MBN-101 in Patients With Moderate to Severe Diabetic Foot Infection (DFI)
Brief Title: A Trial to Assess Safety and Efficacy of Topical MBN-101 in Patients With Moderate/ Severe DFI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Microbion Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MBN-101-202
Record Dates: First submitted 2016-03-11; First posted 2016-03-30 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Foot Infection
MeSH Terms: interventions — 1,2-ethanedithiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MBN-101 (Experimental): MBN-101: a suspension of 150, 375, or 600 microgram (µg)/milliliter (mL) (w:v) BisEDT drug particles in suspension in 3% methylcellulose / 0.5% polysorbate 80 / 10 millimole (mM) sodium chloride / 10 mM sodium phosphate.
  Interventions: Drug: MBN-101
- Vehicle (Placebo Comparator): MBN-101 diluent (placebo): 3% methylcellulose / 0.5% polysorbate 80 / 10 mM sodium chloride / 10 mM sodium phosphate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBN-101 — Topical application
  Other Names: BisEDT
  Arms: MBN-101
Drug: Placebo — Topical application
  Other Names: Vehicle
  Arms: Vehicle

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center study, in patients with moderate to severe diabetic foot infection (DFI), that will be conducted in two parts. In Part I, patients will be enrolled into 1 of 3 escalating dose cohorts at a ratio of 3:1 (Active to Placebo). In Part II, patients will be randomized in a 1:1 ratio (Active to Placebo) based on the optimal dose demonstrated in Part I. Patients will be randomized to receive either topical application of MBN-101 or topical application of vehicle, applied directly to the target site, 3 times per week, for a minimum of 14 days and up to a maximum of 21 days. All patients will also receive systemic antibiotic treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center study that will be conducted in two parts. In Part I, patients will be enrolled into escalating dose cohorts (150, 375, or 600 µg/mL) (N=16/cohort) at a ratio of 3:1 (Active to Placebo). In Part II, patients will be randomized in a 1:1 ratio (Active to Placebo) based on the optimal dose demonstrated in Part I.

Patients with diabetes mellitus and a foot infection with an Infectious Disease Society of America (IDSA) infection severity rating of moderate or severe will be eligible for the trial. Both inpatients and outpatients are eligible if they meet all inclusion/exclusion criteria, however all enrolled patients must remain in-hospital for the first 24 hours after initial dosing. Patients with a need for surgical therapy (e.g., incision and drainage or removal of necrotic tissue) beyond standard bedside wound debridement should not be enrolled.

Patients will be randomized to receive either topical application of MBN-101 or topical application of vehicle, applied directly to the target site, 3 times per week, for a minimum of 14 days and up to a maximum of 21 days. The determination to stop topical antibiotic therapy will be at the discretion of the principal investigator, and should be based on the resolution of findings of infection. All patients will also receive systemic antibiotic treatment based on the protocol defined algorithm. Systemic antibiotic therapy should continue until, but not beyond, the resolution of findings of infection, as outlined in the 2012 IDSA clinical practice guideline for the diagnosis and treatment of diabetic foot infections,

ELIGIBILITY:
Inclusion Criteria:

* Has diabetes mellitus, according to the American Diabetes Association (ADA) criteria
* Has a foot infection as defined by the IDSA guidelines, with a severity rating of moderate or severe
* Either no current or recent (within 72 hours) antibiotic therapy for the DFI,
* Has documented adequate arterial perfusion in the affected limb (either palpable dorsalis pedis or posterior tibial pulses, or normal Doppler wave forms, or a toe blood pressure ≥ 45 mm Hg, or an ankle-brachial index (ABI) of >0.6)

Exclusion Criteria:

* Proven or highly suspected, involvement of bone (i.e., osteomyelitis)
* More than one concurrent, infected, diabetic foot ulcer
* Hemoglobin A1c > 11 on the day of presentation
* Requirement for ongoing immunosuppressive therapy (topical or inhaled corticosteroids are permitted)
* Serum creatinine, alanine aminotransferase (ALT), aspartate aminotransferase (AST) or Alkaline Phosphatase >2 times the upper limit of the normal range of the local testing laboratory
* Absolute neutrophil count <1000
* Any condition that has required treatment with any other bismuth containing compound within the last 2 weeks (i.e., Kaopectate or Pepto-Bismol)
* Participation in an investigational trial to evaluate pharmaceuticals or biologics within the past 3 months
* Need for any surgical therapy beyond debridement to treat the diabetic foot ulcer (e.g., incision and drainage, removal of necrotic tissue)
* Planned lower extremity amputation that will include their infected ulcer
* Known allergy to bismuth and/or MBN-101 excipients (methylcellulose, Tween 80 (polysorbate 80))
* Female patients who are pregnant, lactating, or who have a positive serum human chorionic gonadotropin (pregnancy) as determined by laboratory testing
* Immunocompromised due to illness or organ transplant
* History of any type of cancer (excluding non-melanoma localized skin cancer or completely excised and cured carcinoma-in-situ of uterine cervix)
* History of major medical noncompliance
* Other medical conditions which, in the opinion of the Principal Investigator, would jeopardize the safety of the study subject or impact the validity of the study results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with treatment-related adverse events | From the start of dosing upto 4 weeks following the completion of dosing
  Safety and tolerability will be assessed by treatment-related adverse events
Proportion of participants who are clinically cured | 2 weeks following completion of dosing (up to 5 weeks)
  Clinical cure is defined as the resolution of clinical signs and symptoms of infection 2 weeks following the end of treatment (EOT)

SECONDARY OUTCOMES:
Proportion of participants who are microbiologically cured | 2 weeks following completion of dosing (up to 5 weeks)
  Microbiological cure is defined as the eradication of baseline pathogens 2 weeks following the end of treatment (EOT).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Limb Preservation Platform, Inc, Fresno, California
  - Futuro Clinical Trials, LLC, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipsky BA, Kim PJ, Murphy B, McKernan PA, Armstrong DG, Baker BHJ. Topical pravibismane as adjunctive therapy for moderate or severe diabetic foot infections: A phase 1b randomized, multicenter, double-blind, placebo-controlled trial. Int Wound J. 2024 Apr;21(4):e14817. doi: 10.1111/iwj.14817. PMID 38567778